CLINICAL TRIAL: NCT06009315
Title: Development and Validation for Prognostic Prediction Model of Patients With AcUte Stroke undeRgoing EndOvascular TheRApy (AURORA)
Brief Title: Prognostic Prediction Model of Patients With AcUte Stroke undeRgoing EndOvascular TheRApy (AURORA)
Acronym: AURORA
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor & Director, Beijing Tiantan Hospital
Other Study IDs: LF20230819
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke,; Anesthesia; Predictive Model; Endovascular therapy; Deep learning
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is the leading cause of disability-adjusted life years (DALYs) in China, imposing a heavy burden on society and families. Endovascular therapy (EVT) has opened the 2.0 era of acute ischemic stroke (AIS) treatment, but still up to 1/3 of patients have poor neurological prognosis. The results of several studies at home and abroad and by our team indicate that anesthesia method and perioperative management are one of the key factors affecting the neurological prognosis of EVT treatment in AIS patients. Based on machine learning big data analysis methods, a prognostic model for EVT treatment of AIS patients can be established to guide individualized treatment decisions. Current prediction models only include patients' baseline variables, and lack the inclusion of intraoperative (anesthesia management and interventional process) and postoperative (intensive monitoring treatment) variables, which limits the clinical application of prediction tools. We will establish a large prospective cohort database including preoperative, intraoperative, and postoperative variables, integrate heterogeneous information from multiple sources based on artificial intelligence machine learning algorithms, and build prognostic prediction models with better clinical applicability and calibration, with the aim of optimizing perioperative management of endovascular therapy, guiding individualized clinical decision-making, and improving patients' clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* NIHSS score ≥4;
* Image-confirmed (CTA/MRA/DSA) intracranial large artery occlusion;
* ASPECT (anterior circulation) or PC-ASPECT (posterior circulation) score ≥3;
* Endovascular treatment including arterial thrombolysis, mechanical thrombolysis, and angioplasty (onset to puncture time is recommended to be less than 8 hours for anterior circulation and less than 12 hours for posterior circulation; those exceeding the time window will be determined by the neurointerventionalist through imaging assessment);
* Signed informed consent by the patient or legal representative

Exclusion Criteria:

* Pre-stroke mRS score >2;
* Intracranial bleeding disorders: cerebral hemorrhage, subarachnoid hemorrhage, etc.;
* presence of coagulation disorders, history of systemic bleeding, history of thrombocytopenia or neutropenia;
* Renal insufficiency with elevated blood creatinine (greater than 2 times the upper limit of normal);
* Presence of severe cardiopulmonary disease that, in the opinion of the investigator, makes participation in this study unsuitable; patients with a life expectancy of less than 3 months or otherwise unable to complete this study;
* Contraindication to DSA examination, severe contrast allergy or absolute contraindication to iodine contrast; women of childbearing age who have a negative pregnancy test but refuse to use effective contraception, are pregnant or breast feeding;
* Those who are unable to complete the study due to psychiatric disorders, cognitive or mood disorders;
* Other patients who, in the opinion of the investigator, are not suitable for enrollment in the study (specify reason).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke caused by large undergoing endovascular therapy
Sampling Method: Non-Probability Sample
Enrollment: 949 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence at 90 days | 90±7days after treatment
  modified Rankin Scale of 0-2

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, Liang F, Wu Y, Jia B, Wang A, Zhang X, Zhang K, Hou X, Jian M, Wang Y, Liu H, Miao Z, Han R. Development and Validation of a Two-step Model to Predict Outcomes After Endovascular Treatment for Patients With Acute Ischemic Stroke. J Neurosurg Anesthesiol. 2025 Jul 1;37(3):305-312. doi: 10.1097/ANA.0000000000001008. Epub 2024 Sep 18. PMID 39291867